CLINICAL TRIAL: NCT04178967
Title: A Randomized, Double-blind, Placebo Controlled Trial to Evaluate the Efficacy and Safety of Lebrikizumab in Patients With Moderate to Severe Atopic Dermatitis.
Brief Title: Evaluation of the Efficacy and Safety of Lebrikizumab (LY3650150) in Moderate to Severe Atopic Dermatitis
Acronym: ADvocate2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Dermira, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17802; 2019-002933-12 (EudraCT Number); J2T-DM-KGAC (Other: Eli Lilly and Company); DRM06-AD05 (Other: Dermira, Inc)
Record Dates: First submitted 2019-11-25; First posted 2019-11-26 (Actual); Results first posted 2022-09-16 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases | interventions — lebrikizumab

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, parallel group, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14.
  Maintenance Period (Week 16-Week 52):
  Two placebo SC injections as loading dose on Week 16 and Week 18. One placebo SC injection Q2W until Week 50.
  Interventions: Other: Placebo
- Lebrikizumab Q2W (Experimental): Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
  Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection and one placebo SC injection as maintenance loading dose on Week 16 and Week 18.
  One 250 mg Lebrikizumab SC injection Q2W until Week 50.
  Interventions: Biological: Lebrikizumab
- Lebrikizumab Q4W (Experimental): Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection and one placebo SC injection as maintenance loading dose on Week 16 and two placebo SC injections on Week 18.
  One 250 mg Lebrikizumab SC injection Every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
  Interventions: Biological: Lebrikizumab; Other: Placebo
- Escape Arm (Lebrikizumab Q2W) (Experimental): Maintenance Period (Week 16-Week 52):
  Participants who require topical or systemic rescue treatment for atopic dermatitis during the Induction Period, or are non-responders at Week 16, will be eligible for treatment in an Escape Arm where participants will receive open-label lebrikizumab Q2W from Week 16 through Week 52. In addition, participants who do not maintain an acceptable response during the Maintenance Period (have an EASI score <50% of baseline), will be eligible for the Escape Arm.
  Interventions: Biological: Lebrikizumab

INTERVENTIONS:
Biological: Lebrikizumab — Subcutaneous injection
  Other Names: LY3650150; DRM06
  Arms: Escape Arm (Lebrikizumab Q2W); Lebrikizumab Q2W; Lebrikizumab Q4W
Other: Placebo — Subcutaneous Injection
  Arms: Lebrikizumab Q4W; Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study which is 52 weeks in duration. The study is designed to confirm the safety and efficacy of lebrikizumab as monotherapy for treatment of moderate-to-severe atopic dermatitis utilizing a 16-week induction treatment period and a 36-week long-term maintenance treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults and adolescents (≥12 years and ≥40 kg)
* Chronic atopic dermatitis (according to American Academy of Dermatology Consensus Criteria) that has been present for ≥1 year before the screening visit
* Eczema Area and Severity Index (EASI) score ≥16 at the baseline visit
* Investigator Global Assessment (IGA) score ≥3 (scale of 0 to 4) at the baseline visit
* ≥10% body surface area (BSA) of atopic dermatitis involvement at the baseline visit
* History of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable

Exclusion Criteria:

* Prior treatment with dupilumab or tralokinumab
* Treatment with topical corticosteroids, calcineurin inhibitors or phosphodiesterase-4 inhibitors such as crisaborole within 1 week prior to the baseline visit
* Treatment with any of the following agents within 4 weeks prior to the baseline visit:

  * Immunosuppressive/immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate-mofetil, IFN-γ, Janus kinase inhibitors, azathioprine, methotrexate, etc.)
  * Phototherapy and photochemotherapy (PUVA) for AD
* Treatment with the following prior to the baseline visit:

  * An investigational drug within 8 weeks or within 5 half-lives (if known) of baseline, whichever is longer
  * Cell-depleting biologics, including to rituximab, within 6 months of baseline
  * Other biologics within 5 half-lives (if known) or 16 weeks of baseline, whichever is longer
* Treatment with a live (attenuated) vaccine within 12 weeks of the baseline visit or planned during the study
* Uncontrolled chronic disease that might require bursts of oral corticosteroids, e.g., co-morbid severe uncontrolled asthma
* Evidence of active acute or chronic hepatitis
* History of human immunodeficiency virus (HIV) infection or positive HIV serology
* History of malignancy, including mycosis fungoides, within 5 years before the screening visit, except completely treated in situ carcinoma of the cervix, completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (89):
- United States (40):
  - Investigate MD, Scottsdale, Arizona
  - Northwest Arkansas Clinical Trials Center, Rogers, Arkansas
  - Bakersfield Dermatology and Skin Cancer Medical Group, Bakersfield, California
  - Center For Dermatology Clinical Research, Inc., Fremont, California
  - Woodward Centre, Fresno, California
  - Dermatology Research Associates, Los Angeles, California
  - LA Universal Research Center, INC, Los Angeles, California
  - University Clinical Trials, Inc., San Diego, California
  - San Luis Dermatology & Laser Clinic, San Luis Obispo, California
  - Clinical Physiology Associates, Clinical Study Center, Fort Myers, Florida
  - Direct Helpers Medical Center, Hialeah, Florida
  - The Community Research of South Florida, Hialeah, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Georgia Pollens Clinical Research Centers, Inc, Albany, Georgia
  - Marietta Dermatology Clinical Research, Marietta, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Arlington Dermatology, Rolling Meadows, Illinois
  - NorthShore University HealthSystem, Skokie, Illinois
  - Kansas City Dermatology, PA, Overland Park, Kansas
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - ActivMed Practices and Research, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - Clarkston Skin Research, Clarkston, Michigan
  - Associated Skin Care Specialists, Fridley, Minnesota
  - Central Dermatology PC, St Louis, Missouri
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Dermatology and Skin Surgery Center, Exton, Pennsylvania
  - DermDOX, Hazleton, Pennsylvania
  - Peak Research LLC, Upper Saint Clair, Pennsylvania
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Palmetto Clinical Trial Services, Greenville, South Carolina
  - Arlington Research Center, Inc, Arlington, Texas
  - Innovate Research, LLC, Fort Worth, Texas
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington
- Bulgaria (6):
  - DCC Sveti Georgi, Plovdiv
  - Diagnostic and Consultation Center 14, Sofia
  - Alexandrovska University Hospital, Sofia
  - Euro Derma clinic, Sofia
  - Military Medical Academy, Sofia
  - Medical centre Alitera-Med EOOD, Sofia
- Canada (6):
  - Dr. Chih-ho Hong Medical Inc., Surrey, British Columbia
  - Simcoderm Medical & Surgical Dermatology Centre, Barrie, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - North York Research Inc., North York, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
- Germany (20):
  - Derma-Study-Center Friedrichshafen GmbH, Friedrichshafen, Baden-Wurttemberg
  - Studienzentrum Dr.Beate Schwarz, Langenau, Baden-Wurttemberg
  - Hautarztpraxis am Löwenmarkt, Stuttgart, Baden-Wurttemberg
  - licca Fachklinik, Augsburg, Bavaria
  - Rosenpark Research Geschäftsbereich der Rosenparkklinik GmbH, Darmstadt, Hesse
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Elbe Klinikum Buxtehude, Buxtehude, Lower Saxony
  - Klinische Forschung Osnabrück, Osnabrück, Lower Saxony
  - Fachklinik Bad Bentheim, Bad Bentheim, North Rhine-Westphalia
  - Hautzentrum im Jahrhunderthaus, Bochum, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - SIBAmed Studienzentrum GmbH & Co. KG, Leipzig, Saxony
  - Universität Leipzig - Universitätsklinikum, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein, Lübeck, Schleswig-Holstein
  - Praxis Dr. Michael Dietlen, Augsburg
  - Charité Universitätsmedizin Berlin Campus Buch, Berlin
  - ISA GmbH, Berlin
  - Praxis für Ganzheitliche Dermatologie im Ärztehaus, Berlin
  - Universitätsklinikum Hamburg, Hamburg
  - TFS Trial Form Support GmbH, Hamburg
- Mexico (2):
  - Clinica De Enfermedades Cronicas y Procedimientos Especiales, Morelia, Michoacan Morelia
  - Derma Norte del Bajío, S.C., Aguascalientes
- Singapore (4):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Kk Women'S and Childrens Hospital, Singapore
  - National Skin Centre NSC, Singapore
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Niaosong Dist, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Institutional Review B, Kaohsiung City
  - Taipei Medical University- Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan
- Ukraine (4):
  - Municipal Healthcare Institution Kharkiv City Dermatoverenologic Dispensary N2, Kharkiv
  - Rivne Regional Dermatology and Venereology Dispensary, Rivne
  - Treatment-diagnostic center PE "Asclepius", Uzhhorod
  - Community Institution Zaporizhzhya Regional Dermatovenereology Clinical Hospital of Zaporizhzhya Regional Council, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Sher ER, Golant A, de Bruin-Weller M, Carrascosa JM, Mehta V, Bieber T, Dawson Z, Atwater AR, Zhong J, Rodriguez Calleja L, Boguniewicz M. Lebrikizumab is efficacious in adults and adolescents with moderate-to-severe atopic dermatitis regardless of atopic comorbidities. Ann Allergy Asthma Immunol. 2025 Dec 21:S1081-1206(25)01389-4. doi: 10.1016/j.anai.2025.12.017. Online ahead of print. PMID 41435984
- [Derived] Silverberg JI, Wollenberg A, Stein Gold L, Yosipovitch G, Lio P, Vestergaard C, Stander S, Carrascosa JM, Gallo G, Casillas M, Ding Y, Yang FE, Pierce E, Agell H, Del Rosso J. Lebrikizumab provides stable skin response with no or minimal fluctuations for up to 2 years in patients with atopic dermatitis. Clin Exp Dermatol. 2025 Nov 8:llaf490. doi: 10.1093/ced/llaf490. Online ahead of print. PMID 41206702
- [Derived] Guttman-Yassky E, Sun Z, Mena LR, Hahn N, Nickoloff BJ, Preuss C, Siu K, Natalie CR, Gallo G, Wolf E, Eyerich K, Aparici M, Benschop RJ, Okragly A. Lebrikizumab Rapidly Lowers Inflammatory Biomarkers with Clinical Correlations in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2025 Sep;15(9):2595-2614. doi: 10.1007/s13555-025-01481-4. Epub 2025 Jul 15. PMID 40663228
- [Derived] Simpson E, Fernandez-Penas P, de Bruin-Weller M, Lio PA, Chu CY, Ezzedine K, Agell H, Casillas M, Ding Y, Yang FE, Pierce E, Bieber T. Improvement Across Dimensions of Disease with Lebrikizumab Use in Atopic Dermatitis: Two Phase 3, Randomized, Double-Blind, Placebo-Controlled Monotherapy Trials (ADvocate1 and ADvocate2). Adv Ther. 2025 Jan;42(1):132-143. doi: 10.1007/s12325-024-02974-y. Epub 2024 Sep 9. PMID 39249591
- [Derived] Silverberg JI, Wollenberg A, Stein Gold L, Del Rosso J, Yosipovitch G, Lio P, Carrascosa JM, Gallo G, Ding Y, Xu Z, Casillas M, Pierce E, Agell H, Stander S. Patients with Moderate-to-Severe Atopic Dermatitis Maintain Stable Response with No or Minimal Fluctuations with 1 Year of Lebrikizumab Treatment. Dermatol Ther (Heidelb). 2024 Aug;14(8):2249-2260. doi: 10.1007/s13555-024-01226-9. Epub 2024 Aug 10. PMID 39123054
- [Derived] Yosipovitch G, Lio P, Legat FJ, Chovatiya R, Deleuran M, Pierce E, Casillas M, Ding Y, Yang FE, Bardolet L, Stander S. Stable Response and Sustained Improvement of Itch and Sleep Symptoms in Patients with Atopic Dermatitis Treated with Lebrikizumab over 52 Weeks. Dermatol Ther (Heidelb). 2024 Aug;14(8):2171-2180. doi: 10.1007/s13555-024-01225-w. Epub 2024 Jul 13. PMID 39002092
- [Derived] Lio PA, Armstrong A, Gutermuth J, Nosbaum A, Sofen H, Gil EG, Casillas M, Chen S, Sun L, Pierce E, Elmaraghy H, Dawson Z, Torres T. Lebrikizumab Improves Quality of Life and Patient-Reported Symptoms of Anxiety and Depression in Patients with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1929-1943. doi: 10.1007/s13555-024-01199-9. Epub 2024 Jun 26. PMID 38922484
- [Derived] Simpson EL, de Bruin-Weller M, Hong HC, Staumont-Salle D, Blauvelt A, Eyerich K, Gooderham M, Shahriari M, Mallbris L, Atwater AR, Rueda MJ, Ding Y, Liu Z, Agell H, Silverberg JI. Lebrikizumab Provides Rapid Clinical Responses Across All Eczema Area and Severity Index Body Regions and Clinical Signs in Adolescents and Adults with Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 May;14(5):1145-1160. doi: 10.1007/s13555-024-01158-4. Epub 2024 May 3. PMID 38700646
- [Derived] Soung J, Stander S, Gutermuth J, Pau-Charles I, Dawson Z, Yang FE, Sun L, Pierce E, Elmaraghy H, Stein-Gold L. Lebrikizumab monotherapy impacts on quality of life scores through improved itch and sleep interference in two Phase 3 trials. J Dermatolog Treat. 2024 Dec;35(1):2329240. doi: 10.1080/09546634.2024.2329240. Epub 2024 Apr 28. PMID 38679419
- [Derived] Blauvelt A, Thyssen JP, Guttman-Yassky E, Bieber T, Serra-Baldrich E, Simpson E, Rosmarin D, Elmaraghy H, Meskimen E, Natalie CR, Liu Z, Xu C, Pierce E, Morgan-Cox M, Garcia Gil E, Silverberg JI. Efficacy and safety of lebrikizumab in moderate-to-severe atopic dermatitis: 52-week results of two randomized double-blinded placebo-controlled phase III trials. Br J Dermatol. 2023 May 24;188(6):740-748. doi: 10.1093/bjd/ljad022. PMID 36994947
- [Derived] Silverberg JI, Guttman-Yassky E, Thaci D, Irvine AD, Stein Gold L, Blauvelt A, Simpson EL, Chu CY, Liu Z, Gontijo Lima R, Pillai SG, Seneschal J; ADvocate1 and ADvocate2 Investigators. Two Phase 3 Trials of Lebrikizumab for Moderate-to-Severe Atopic Dermatitis. N Engl J Med. 2023 Mar 23;388(12):1080-1091. doi: 10.1056/NEJMoa2206714. Epub 2023 Mar 15. PMID 36920778
- See also: Evaluation of the Efficacy and Safety of Lebrikizumab (LY3650150) in Moderate to Severe Atopic Dermatitis (ADvocate2) — https://trials.lillytrialguide.com/en-US/trial/AmPN68cQaViDZ8pT3j6hD

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During the Induction period (16-weeks): Participants were randomly assigned to either 250 mg lebrikizumab Q2W or placebo; At week 16, participants who responded to treatment, defined as having an Investigator Global Assessment (IGA) of 0 or 1 or a 75% reduction in Eczema Area and Severity Index (EASI-75) from Baseline to Week 16 entered Maintenance Period and were re-randomized (2:2:1) to: lebrikizumab 250 mg Q2W, lebrikizumab 250 mg Q4W, or placebo (Continued)
Pre-assignment Details: (Continued) Induction non-responder (i.e.) participants who do not achieve an IGA of 0 or 1 or an EASI-75 at Week 16 and maintenance non-responders (i.e.) those not maintaining an EASI-50 response at week 24, 32, 40, and 48 following week 16 re-randomization were assigned to an Escape Arm and received lebrikizumab 250 mg as open-label treatment Q2W through Week 52.
Groups:
- Induction - Placebo: Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14.
- Induction - Lebrikizumab Q2W: Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
- Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO): Maintenance Secondary Population: Maintenance Period (Week 16 to Week 52):
  One SC injection of Placebo Q2W until Week 50. Two placebo SC injections as loading dose on Week 16 and Week 18.
- Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W: Maintenance Secondary Population: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
  For participants who received placebo in the Induction Period, the maintenance loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16. Two placebo injections on Week 18.
- Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W: Maintenance Secondary Population: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection Q2W until Week 50.
  For participants who received placebo in the Induction Period, the maintenance loading dose is:
  Two 250 mg Lebrikizumab SC injections on Week 16. Two 250 mg Lebrikizumab SC injections on Week 18.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo: Maintenance Primary Population: Maintenance Period (Week 16 to Week 52): One SC injection of Placebo Q2W until Week 50.
  Two placebo SC injections as loading dose on Week 16 and Week 18.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W: Maintenance Primary Population: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
  To maintain the blind, for participants who received Lebrikizumab in the Induction Period, the maintenance loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16. Two placebo injections on Week 18.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W: Maintenance Primary Population: Maintenance Period (Week 16 to Week 52):
  One 250 mg Lebrikizumab SC injection Q2W until Week 50.
  To maintain the blind, for participants who received Lebrikizumab in the Induction Period, the maintenance loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 16. One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 18.
- Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W: Maintenance Escape Period (Week 16 to Week 52):
  Blinded loading doses based on prior treatment assignment will be administered, followed by one 250 mg Lebrikizumab SC injection Q2W until Week 50 in an open-label fashion.
  For participants who received placebo in the Induction Period, the loading dose is:
  Two 250 mg Lebrikizumab SC injection on Week 16. Two 250 mg Lebrikizumab SC injections on Week 18.
  For participants who do not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses will be administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
  Participants who did not achieve an EASI-50 response after 8 weeks in the Escape Arm were terminated from the study.
- Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W: Maintenance Escape Period (Week 16 to Week 52):
  Blinded loading doses based on prior treatment assignment will be administered, followed by one 250 mg Lebrikizumab SC injection Q2W until Week 50 in an open-label fashion.
  To maintain the loading dose blind, for participants who received Lebrikizumab in the Induction Period, the loading dose is:
  One 250 mg Lebrikizumab SC injection and one placebo on Week16. One 250 mg Lebrikizumab SC injection and one placebo SC injection on Week 18.
  For participants who do not maintain an acceptable response during the Maintenance Period and entered the Escape Arm, the loading doses will be administrated at entry and 2 weeks after entry based on the treatment assignment prior to entering escape arm.
  Participants who did not achieve an EASI-50 response after 8 weeks in the Escape Arm were terminated from the study.
- Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W: Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W.
Period: Induction Period
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO) | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W
Started | 150 | 295 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 149 | 295 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 133 (Completed includes Responders n=25; Non responders n=108) | 273 (Completed includes Responders n=148; Non responders n=125) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 17 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Due to Epidemic/Pandemic | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 4 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Missed Study Visits | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Maintenance Blinded Treatment Period
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO) | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W
Started | 0 (Participants were assigned to this arm only during Induction Period.) | 0 (Participants were assigned to this arm only during Induction Period.) | 5 (Only those participants who responded to induction placebo or Lebrikizumab at week 16 entered the Maintenance Period.) | 9 (Only those participants who responded to induction placebo or Lebrikizumab at week 16 entered the Maintenance Period.) | 11 (Only those participants who responded to induction placebo or Lebrikizumab at week 16 entered the Maintenance Period.) | 30 (Only those participants who responded to induction placebo or Lebrikizumab at week 16 entered the Maintenance Period.) | 59 (Only those participants who responded to induction placebo or Lebrikizumab at week 16 entered the Maintenance Period.) | 59 (Only those participants who responded to induction placebo or Lebrikizumab at week 16 entered the Maintenance Period.) | 0 | 0 | 0
Received at Least One Dose of Study Drug | 0 | 0 | 5 | 9 | 11 | 30 | 59 | 59 | 0 | 0 | 0
Completed | 0 | 0 | 4 | 6 | 9 | 22 | 51 | 42 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 3 | 2 | 8 | 8 | 17 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 4 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 1 | 1 | 1 | 1 | 4 | 6 | 0 | 0 | 0
Not completed — Entered Escape Arm | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 6 | 0 | 0 | 0
Period: Maintenance Open Label Escape Arm
Arm/Group | Induction - Placebo | Induction - Lebrikizumab Q2W | Maintenance Blinded Treatment - Placebo Responder/Placebo (PBO) | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Placebo Responder/Lebrikizumab 250 Q2W | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Placebo Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 16 - Maintenance Open Label - Lebrikizumab Nonresponder/ Lebrikizumab 250 Q2W | Escape Arm Week 24 to 48 - Maintenance Open Label Lebrikizumab 250 Q2W
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108 (Only those participants who did not respond to induction placebo or Lebrikizumab entered Escape Arm at week 16.) | 125 (Only those participants who did not respond to induction placebo or Lebrikizumab entered Escape Arm at week 16.) | 11 (Only those participants who did not respond to treatment during maintenance period (i.e.) not maintaining an EASI-50 response at Weeks 24, 32, 40, or 48 were entered.)
Received at Least One Dose of Study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 108 | 125 | 11
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 85 | 83 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 23 | 42 | 3
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 27 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 9 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Participant Missed Study Visits | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol.
Groups:
- Placebo: Induction Period (Baseline-Week 16):
  Two subcutaneous (SC) injections of Placebo as a loading dose at Baseline and Week 2 followed by a single injection every 2 weeks (Q2W) from Week 4 until Week 14.
- Lebrikizumab Q2W: Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lebrikizumab Q2W | Total
Number analyzed (Participants) | 150 | 295 | 445
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 33 | 50
  Between 18 and 65 years | 123 | 239 | 362
  >=65 years | 10 | 23 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (17.15) | 36.5 (16.64) | 36.2 (16.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 147 | 226
  Male | 71 | 148 | 219
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 44 | 78 | 122
  Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
  Black or African American | 10 | 26 | 36
  White | 89 | 181 | 270
  More than one race | 3 | 4 | 7
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 16 | 42 | 58
  Singapore | 8 | 11 | 19
  United States | 64 | 121 | 185
  Taiwan | 21 | 39 | 60
  Ukraine | 3 | 8 | 11
  Mexico | 3 | 6 | 9
  Bulgaria | 7 | 15 | 22
  Germany | 28 | 53 | 81

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Investigator Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their atopic dermatitis (AD), based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to Good Clinical Practice (GCP) issues. Markov Chain Monte Carlo Multiple Imputation (MCMC-MI) was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 10.8 [5.7 to 15.9] | 33.2 [27.5 to 38.9]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000004, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.9, 95% CI 2-sided [14.2 to 29.6]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area And Severity Index (EASI-75) (≥75% Reduction in EASI Score) From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% reduction from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: All randomized participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 18.1 [11.7 to 24.5] | 52.1 [46.1 to 58.0]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 33.3, 95% CI 2-sided [24.4 to 42.2]

3. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 2
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on an overall assessment of the degree of erythema, papulation/induration, oozing/crusting, and lichenification.
Time Frame: Baseline to Week 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 0 [0.0 to 0.0] | 0.7 [-0.3 to 1.7]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.308463, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.7, 95% CI 2-sided [-0.3 to 1.7]

4. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 4
Description: as for outcome 3
Time Frame: Baseline to Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 1.4 [0.0 to 3.3] | 9.0 [5.6 to 12.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.001607, Cochran-Mantel-Haenszel; Risk Difference (RD) = 8.1, 95% CI 2-sided [4.1 to 12.0]

5. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16
Description: as for outcome 3
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 10.8 [5.7 to 15.9] | 33.2 [27.5 to 38.9]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000004, Cochran-Mantel-Haenszel; Risk Difference (RD) = 21.9, 95% CI 2-sided [14.2 to 29.6]

6. Secondary Outcome: Percentage of Participants Achieving EASI-90 (≥90% Reduction in EASI Score) From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  The EASI-90 responder is defined as a participant who achieves a ≥ 90% reduction from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 9.5 [4.6 to 14.3] | 30.7 [25.2 to 36.2]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000008, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.7, 95% CI 2-sided [13.3 to 28.1]

7. Secondary Outcome: Percentage Change in Pruritus Numerical Rating Scale (NRS) Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Least Squares (LS) Mean was calculated using analysis of covariance (ANCOVA) model with treatment and randomization strata (region, disease severity, age) as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with a Baseline Pruritus NRS score >0, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: percentage change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage change | -9.02 (3.868) | -36.56 (3.321)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -27.53, 95% CI 2-sided [-34.9 to -20.2]

8. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4-points at Baseline Who Achieve a ≥4-point Reduction in Pruritus NRS Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline to Week 16
Population: All randomized participants, with a Baseline Pruritus NRS score ≥4, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 134 | 253
percentage of participants | 11.5 [6.0 to 16.9] | 39.8 [33.6 to 46.0]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 28.3, 95% CI 2-sided [20.0 to 36.5]

9. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5-points at Baseline Who Achieve a ≥4-point Reduction in Pruritus NRS Score From Baseline to Week 16
Description: as for outcome 8
Time Frame: Baseline to Week 16
Population: All randomized participants, with Baseline Pruritus NRS score ≥ 5, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 122 | 234
percentage of participants | 11.8 [6.0 to 17.6] | 41.6 [35.1 to 48.1]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 29.7, 95% CI 2-sided [21.0 to 38.4]

10. Secondary Outcome: Percentage Change in EASI Score From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
  LS Mean was calculated using ANCOVA model with treatment, stratification factors of geographic region, age group, baseline IGA score (IGA 3 versus 4) as fixed factors baseline value as covariate.
Time Frame: Baseline, Week 16
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percent change | -27.96 (3.893) | -61.53 (3.300)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -33.57, 95% CI 2-sided [-41.2 to -26.0]

11. Secondary Outcome: Change From Baseline in Percent Body Surface Area (BSA) at Week 16
Description: The BSA affected by AD will be assessed for 4 separate body regions: head and neck, trunk (including genital region), upper extremities, and lower extremities (including the buttocks). Each body region will be assessed for disease extent ranging from 0% to 100% involvement. BSA was calculated using the participant's palm using the 1% rule, 1 palm was equivalent to 1% with estimates of the number of palms it takes to cover the affected AD area. Maximum number of palms were 10 palms for head and neck (10%), 20 palms for upper extremities (20%), 30 palms for trunk, including axilla and groin (30%), 40 palms for lower extremities, including buttocks (40%). Percent of BSA for a body region was calculated as = total number of palms in a body region * % surface area equivalent to 1 palm. Overall percent BSA of all 4 body regions ranges from 0% to 100 % with higher values representing greater severity of AD.
Time Frame: Baseline, Week 16
Population: All randomized participants, with observed BSA data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. The MMRM included treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit, geographic region, age group, baseline IGA score.
Measure: Least Squares Mean (Standard Error); unit: percentage of BSA
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 77 | 213
percentage of BSA | -14.0 (1.94) | -30.2 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Mixed Models Analysis; LS Mean Difference (Final Values) = -16.2, 95% CI 2-sided [-20.3 to -12.0]

12. Secondary Outcome: Percentage of Participants Achieving EASI-90 From Baseline to Week 4
Description: as for outcome 6
Time Frame: Baseline to Week 4
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percentage of participants | 1.5 [-0.5 to 3.5] | 6.3 [3.4 to 9.2]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.022921, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.9, 95% CI 2-sided [1.4 to 8.4]

13. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 16
Description: The DLQI is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
  LS Mean was calculated using the ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing baseline DLQI score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 118 | 218
score on a scale | -2.4 (1.17) | -7.3 (1.16)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -4.9, 95% CI 2-sided [-6.3 to -3.5]

14. Secondary Outcome: Percentage of Participants Achieving ≥4-point Improvement in DLQI From Baseline to Week 16
Description: The DLQI is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms, embarrassment, shopping and home care, clothes, social and leisure, sport, work or study, close relationships, sex, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
Time Frame: Baseline to Week 16
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 118 | 218
percentage of participants | 32.8 [24.1 to 41.4] | 65.4 [59.0 to 71.9]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 32.9, 95% CI 2-sided [22.2 to 43.6]

15. Secondary Outcome: Percentage of Participants With a DLQI Total Score of ≥4-point at Baseline Achieving ≥4-point Improvement in DLQI From Baseline to Week 16
Description: as for outcome 14
Time Frame: Baseline to Week 16
Population: All randomized participants, with a DLQI Total Score of ≥4-point at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 115 | 215
percentage of participants | 33.6 [24.8 to 42.5] | 66.3 [59.9 to 72.8]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000001, Cochran-Mantel-Haenszel; Risk Difference (RD) = 33.0, 95% CI 2-sided [22.2 to 43.8]

16. Secondary Outcome: Percentage Change in Sleep-loss Score From Baseline to Week 16
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary. LS Mean was calculated using ANCOVA model with treatment, baseline value, and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized participants, with baseline sleep-loss score >0, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percent change | -11.29 (5.393) | -48.37 (4.590)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -37.09, 95% CI 2-sided [-47.4 to -26.8]

17. Secondary Outcome: Change From Baseline in Sleep-loss Score at Week 16
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing baseline Sleep-loss score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
score on a scale | -0.35 (0.095) | -1.05 (0.080)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-0.9 to -0.5]

18. Secondary Outcome: Percentage of Participants With a Sleep-loss Score ≥2 Points at Baseline Who Achieve a ≥2 Points Reduction From Baseline to Week 16
Description: Sleep Loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all)]. Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant using an electronic diary.
Time Frame: Baseline to Week 16
Population: All randomized participants, with baseline sleep-loss score ≥2 Points, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 97 | 161
percentage of participants | 8.2 [2.5 to 13.9] | 28.0 [21.0 to 35.0]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000571, Cochran-Mantel-Haenszel; Risk Difference (RD) = 18.9, 95% CI 2-sided [9.6 to 28.1]

19. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 1
Description: as for outcome 8
Time Frame: Baseline to Week 1
Population: All randomized participants, with a Pruritus NRS Score of ≥4 Points at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 134 | 253
percentage of participants | 0.0 [0.0 to 0.0] | 0.4 [0.0 to 1.2]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.469221, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.4, 95% CI 2-sided [-0.4 to 1.2]

20. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 8
Time Frame: Baseline to Week 2
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 134 | 253
percentage of participants | 0.7 [0.0 to 2.2] | 3.6 [1.3 to 5.9]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.113194, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.7, 95% CI 2-sided [-0.1 to 5.4]

21. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥4 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 4
Description: as for outcome 8
Time Frame: Baseline to Week 4
Population: as for outcome 19
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 134 | 253
percentage of participants | 3.0 [0.1 to 6.0] | 16.8 [12.2 to 21.4]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000230, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.2, 95% CI 2-sided [7.7 to 18.7]

22. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 1
Description: as for outcome 8
Time Frame: Baseline to Week 1
Population: All randomized participants, with a Pruritus NRS Score of ≥5 Points at Baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MCMC-MI was used to handle missing data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 122 | 234
percentage of participants | 0.0 [0.0 to 0.0] | 0.4 [0.0 to 1.3]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.468160, Cochran-Mantel-Haenszel; Risk Difference (RD) = 0.4, 95% CI 2-sided [-0.4 to 1.3]

23. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 2
Description: as for outcome 8
Time Frame: Baseline to Week 2
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 122 | 234
percentage of participants | 0.8 [0.0 to 2.4] | 3.9 [1.4 to 6.3]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.115770, Cochran-Mantel-Haenszel; Risk Difference (RD) = 2.9, 95% CI 2-sided [-0.1 to 5.8]

24. Secondary Outcome: Percentage of Participants With a Pruritus NRS Score of ≥5 Points at Baseline Who Achieve a ≥4-point Reduction From Baseline to Week 4
Description: as for outcome 8
Time Frame: Baseline to Week 4
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 122 | 234
percentage of participants | 3.3 [0.1 to 6.6] | 18.1 [13.2 to 23.1]
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000252, Cochran-Mantel-Haenszel; Risk Difference (RD) = 14.2, 95% CI 2-sided [8.2 to 20.1]

25. Secondary Outcome: Percentage Change in SCORing Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: SCORAD is validated tool for assessing the extent and intensity of AD, it consists of 3 components: A=extent of AD as a percentage of each defined body area and reported as sum of all areas, with maximum score of 100%. B=severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) assessed using following scale: none=0, mild=1, moderate=2, or severe=3 for maximum of 18 total points. C=subjective assessment of itch and sleeplessness recorded by participant on visual analog scale (VAS), where 0=no itch/no sleeplessness and 10=worst imaginable itch/sleeplessness with maximum score of 20. SCORAD total score is calculated: A/5+7*B/2+ C to give total score range of 0 to 103, where 0=no disease to 103=severe disease. LS Mean was calculated using ANCOVA model with treatment group and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with baseline SCORAD >0, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing Values were imputed using last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
percent change | -13.81 (3.197) | -44.57 (2.677)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, ANCOVA; LS Mean Difference (Final Values) = -30.76, 95% CI 2-sided [-36.93 to -24.59]

26. Secondary Outcome: Pharmacokinetics (PK): Trough Serum Concentrations of Lebrikizumab in Maintenance Period (C-trough)
Description: C-trough was the concentration of study drug in the blood immediately before the next dose was administered. Trough serum concentration of Lebrikizumab was assessed at predose week 52.
Time Frame: Predose at Week 52
Population: All participants who received 250 mg Q2W or 250 mg Q4W in the Maintenance Period and had evaluable PK data at Week 52. The 250 mg Q2W PK population also includes participants from the Escape Arm (Induction period non-responders and Maintenance Period non-responders who received open-label 250 mg Q2W dosing).
Measure: Mean (Standard Deviation); unit: micrograms/milliliter (µg/mL)
Groups:
- Maintenance 250 mg Lebrikizumab Q4W: 250 mg Lebrikizumab administered SC injection Q4W.
- Maintenance 250 mg Lebrikizumab Q2W and 250 mg Lebrikizumab Escape Q2W: 250 mg Lebrikizumab administered SC injection Q2W.
Arm/Group | Maintenance 250 mg Lebrikizumab Q4W | Maintenance 250 mg Lebrikizumab Q2W and 250 mg Lebrikizumab Escape Q2W
Number analyzed (Participants) | 51 | 206
micrograms/milliliter (µg/mL) | 46.7 (24.8) | 90.5 (40.1)

27. Secondary Outcome: Percentage of Participants From Those Re-randomized Having Achieved EASI-75 at Week 16 Who Continue to Exhibit EASI-75 at Week 52 (EASI-75 Calculated Relative to Baseline EASI Score)
Description: The EASI assesses objective physician estimates of 2 dimensions of AD - disease extent, i.e., percentage of skin affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI-75 score was obtained by weight-averaging these 4 scores and will range from 0 (none) to 72 (severe).
  The EASI-75 responder is defined as a participant who achieves a ≥ 75% reduction from baseline in the EASI score.
Time Frame: Baseline to Week 52
Population: All participants who were randomized to Lebrikizumab 250 mg Q2W at Baseline Visit and re-randomized to Lebrikizumab 250 mg Q2W, Lebrikizumab 250 mg Q4W or placebo at Week 16 and received at least 1 dose of study treatment during the maintenance period and had evaluable EASI-75 data at week 52.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo: Participants received placebo administered SC injection Q2W
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W: Participants received 250 mg Lebrikizumab administered SC injection Q4W.
- Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W: Participants received 250 mg Lebrikizumab administered SC injection Q2W.
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 27 | 53 | 51
percentage of participants | 72.0 [53.0 to 91.0] | 84.7 [73.0 to 96.4] | 77.4 [65.4 to 89.4]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.238245, Cochran-Mantel-Haenszel; Risk Difference (RD) = 12.8, 95% CI 2-sided [-9.5 to 35.1]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.612427, Cochran-Mantel-Haenszel; Risk Difference (RD) = 4.8, 95% CI 2-sided [-17.8 to 27.3]

28. Secondary Outcome: Percentage of Participants From Those Re-randomized Having Achieved IGA 0 or 1 and a ≥2-point Improvement From Baseline at Week 16 Who Continue to Exhibit an IGA 0 or 1 and a ≥2-point Improvement From Baseline at Week 52
Description: as for outcome 3
Time Frame: Baseline to Week 52
Population: All participants who were randomized to Lebrikizumab 250 mg Q2W at Baseline Visit and re-randomized to Lebrikizumab 250 mg Q2W, Lebrikizumab 250 mg Q4W or placebo at Week 16 and received at least 1 dose of study treatment during the maintenance period and had evaluable IGA data at week 52.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 16 | 32 | 32
percentage of participants | 49.8 [23.7 to 75.8] | 80.6 [65.9 to 95.3] | 64.6 [47.2 to 82.0]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.033876, Cochran-Mantel-Haenszel; Risk Difference (RD) = 32.6, 95% CI 2-sided [2.6 to 62.5]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.407417, Cochran-Mantel-Haenszel; Risk Difference (RD) = 13.4, 95% CI 2-sided [-17.5 to 44.3]

29. Secondary Outcome: Percentage of Participants From Those With a Pruritus NRS of ≥4-points at Baseline Re-randomized Having Achieved ≥4-point Reduction From Baseline at Week 16 Who Continue to Exhibit ≥4-point Reduction From Baseline at Week 52
Description: as for outcome 8
Time Frame: Baseline to Week 52
Population: All participants who were randomized to Lebrikizumab 250 mg Q2W at Baseline Visit and re-randomized to Lebrikizumab 250 mg Q2W, Lebrikizumab 250 mg Q4W or placebo at Week 16 and received at least 1 dose of study treatment during the maintenance period and had evaluable data at week 52.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 11 | 36 | 23
percentage of participants | 67.6 [38.6 to 96.7] | 88.1 [77.1 to 99.1] | 90.3 [77.3 to 103.2]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.159281, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.3, 95% CI 2-sided [-11.4 to 52.0]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.164950, Cochran-Mantel-Haenszel; Risk Difference (RD) = 20.4, 95% CI 2-sided [-10.6 to 51.4]

30. Secondary Outcome: Percentage of Participants From Those With a Pruritus NRS of ≥5-points at Baseline Re-randomized Having Achieved ≥4-point Reduction From Baseline at Week 16 Who Continue to Exhibit ≥4-point Reduction From Baseline at Week 52
Description: as for outcome 8
Time Frame: Baseline to Week 52
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: percentage of partcipants
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 11 | 34 | 22
percentage of partcipants | 67.6 [38.6 to 96.7] | 87.4 [75.8 to 99.0] | 94.4 [83.6 to 105.1]
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.179704, Cochran-Mantel-Haenszel; Risk Difference (RD) = 19.7, 95% CI 2-sided [-12.2 to 51.2]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.083080, Cochran-Mantel-Haenszel; Risk Difference (RD) = 24.3, 95% CI 2-sided [-6.5 to 55.1]

31. Secondary Outcome: Percentage Change in SCORAD (From Those Re-randomized Having Achieved EASI-75 at Week 16) From Baseline at Week 52
Description: SCORAD is a validated tool for assessing the extent and intensity of AD, it consists of 3 components: A=extent of AD as a percentage of each defined body area and reported as sum of all areas, with maximum score of 100%. B=severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) assessed using following scale: none=0, mild=1, moderate=2, or severe=3 for maximum of 18 total points. C=subjective assessment of itch and sleeplessness recorded by participant on VAS, where 0=no itch/no sleeplessness and 10=worst imaginable itch/sleeplessness with maximum score of 20. SCORAD total score is calculated: A/5+7*B/2+ C to give total score range of 0 to 103, where 0=no disease to 103=severe disease. LS Mean was calculated using ANCOVA model with treatment group and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 52
Population: All participants who were randomized to Lebrikizumab 250 mg Q2W at Baseline Visit and re-randomized to Lebrikizumab 250 mg Q2W, Lebrikizumab 250 mg Q4W or placebo at Week 16 and received at least 1 dose of study treatment during the maintenance period and had evaluable data at week 52. Missing Values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W | Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W
Number analyzed (Participants) | 27 | 53 | 51
percent change | -67.60 (3.767) | -73.89 (2.718) | -73.85 (2.764)
Statistical Analysis 1: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q4W; Test type: Superiority; p = 0.176748, ANCOVA; LS Mean Difference (Final Values) = -6.29, 95% CI 2-sided [-15.46 to 2.87]
Statistical Analysis 2: Comparison: Maintenance Blinded Treatment - Lebrikizumab Responder/Placebo vs Maintenance Blinded Treatment - Lebrikizumab Responder/Lebrikizumab 250 Q2W; Test type: Superiority; p = 0.183151, ANCOVA; LS Mean Difference (Final Values) = -6.25, 95% CI 2-sided [-15.48 to 2.99]

32. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) at Week 16 - Health State Index
Description: The European Quality of Life-5 Dimensions-5 Level (EQ-5D-5L) is a is a 2-part questionnaire which measure health status of the participant. The first component (Health state) is a descriptive system of the respondent's health comprised of the following 5 participant-reported dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The responses are used to derive the health state index scores using the United Kingdom (UK) algorithm, with scores ranging from -0.594 to 1, and the United States (US) algorithm, with scores ranging from -0.109 to 1. A higher score indicates better health state.
  LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing EQ-5D-5L- Health State Index data at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing Values were imputed using last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 146 | 281
score on a scale
  Health State Index UK | 0.0 (0.02) | 0.1 (0.02)
  Health State Index US | 0.0 (0.01) | 0.1 (0.01)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; UK; Test type: Superiority; p = 0.000001, ANCOVA; LS Mean Difference (Final Values) = 0.1, 95% CI 2-sided [0.1 to 0.1]
Statistical Analysis 2: Comparison: Placebo vs Lebrikizumab Q2W; US; Test type: Superiority; p = 0.000001, ANCOVA; LS Mean Difference (Final Values) = 0.1, 95% CI 2-sided [0.0 to 0.1]

33. Secondary Outcome: Change From Baseline in EQ-5D-5L at Week 16 - Visual Analog Scale (VAS)
Description: The EQ-5D-5L is a 2-part measurement. The second part is assessed using a VAS that ranged from 0 to 100 millimeter (mm), where 0 is the worst health you can imagine and 100 is the best health you can imagine. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing EQ-5D-5L-VAS data at baseline, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: millimeters (mm)
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 145 | 277
millimeters (mm) | 5.2 (1.62) | 9.7 (1.36)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.005304, ANCOVA; LS Mean Difference (Final Values) = 4.5, 95% CI 2-sided [1.3 to 7.6]

34. Secondary Outcome: Change From Baseline in Patient Oriented Eczema Measure (POEM) at Week 16
Description: POEM is a 7-item, validated, questionnaire used by the participant to assess disease symptoms over the last week. The participant is asked to respond to 7 questions on skin dryness, itching, flaking, cracking, sleep loss, bleeding and weeping. All 7 answers carry equal weight with a total possible score from 0 to 28 (answers scored as: No days=0; 1-2 days = 1; 3-4 days = 2; 5-6 days = 3; everyday = 4). A high score is indicative of a poor quality of life. POEM responses will be captured using an electronic diary and transferred into the clinical database. LS Mean was calculated using MMRM model using treatment, baseline value, visit, the interaction of the baseline value-by-visit, the interaction of treatment by-visit as covariates, geographic region, age group, baseline IGA (3 versus 4) score as fixed.
Time Frame: Baseline, Week 16
Population: All randomized participants, with observed POEM data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MMRM was used to handle all missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 65 | 184
score on a scale | -3.5 (0.77) | -9.5 (0.52)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p < 0.000001, Mixed Models Analysis; LS Mean Difference (Final Values) = -6.0, 95% CI 2-sided [-7.7 to -4.3]

35. Secondary Outcome: Change From Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety at Week 16-Adolescents
Description: PROMIS® is a set of person-centered measures that evaluates and monitors physical, mental, and social health in adults and children. Participants ≤17 years will complete pediatric versions for the duration of the study. PROMIS anxiety has 8 questions on Emotion Distress-Anxiety (or Pediatric Anxiety Symptom). Each question has 5 response options with values from 1 to 5. Total raw scores were converted to T-Scores (mean = 50 and a standard deviation = 10) with higher scores representing greater anxiety. LS Mean was calculated using the ANCOVA model with treatment and stratification factors of geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized, adolescent participants, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 17 | 30
T-score | 0.12 (2.129) | -2.79 (1.550)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.241275, ANCOVA; LS Mean Difference (Final Values) = -2.91, 95% CI 2-sided [-7.85 to 2.03]

36. Secondary Outcome: Change From Baseline in PROMIS Anxiety at Week 16 - Adults
Description: as for outcome 35
Time Frame: Baseline, Week 16
Population: All randomized, adults participants, with Week 16 PROMIS anxiety data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing Values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 128 | 246
T-score | -0.45 (0.580) | -3.18 (0.422)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000116, ANCOVA; LS Mean Difference (Final Values) = -2.74, 95% CI 2-sided [-4.12 to -1.36]

37. Secondary Outcome: Change From Baseline in PROMIS Depression at Week 16- Adolescents
Description: as for outcome 35
Time Frame: Baseline, Week 16
Population: as for outcome 35
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 17 | 30
T-score | -0.57 (2.047) | -1.67 (1.493)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.645132, ANCOVA; LS Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-5.86 to 3.67]

38. Secondary Outcome: Change From Baseline in PROMIS Depression at Week 16- Adults
Description: as for outcome 35
Time Frame: Baseline, Week 16
Population: All randomized, adult participants, with Week 16 PROMIS Depression data, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 128 | 246
T-score | 0.16 (0.540) | -2.59 (0.392)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.000031, ANCOVA; LS Mean Difference (Final Values) = -2.75, 95% CI 2-sided [-4.03 to -1.47]

39. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) Score at Week 16 in Participants Who Have Self-reported Comorbid Asthma
Description: The ACQ-5 is a five-item, self-completed questionnaire, which is used as a measure of asthma control of a participant. The five questions (concerning nocturnal awakening, waking in the morning, activity limitation, shortness of breath and wheeze) enquire about the frequency and/or severity of symptoms over the previous week. The response options for all these questions range from zero (no impairment/limitation) to six (total impairment/ limitation) scale. The ACQ-5 score is the average of the individual item scores and ranges from 0 (totally controlled) to 6 (severely uncontrolled). Higher scores indicate lower asthma control.
  LS Mean was calculated using ANCOVA with treatment, geographic region, age group, baseline IGA (3 versus 4) score as fixed factors and baseline value as covariate.
Time Frame: Baseline, Week 16
Population: All randomized participants, with non-missing baseline ACQ-5 score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. Missing values were imputed using LOCF method.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 35 | 75
score on a scale | 0.19 (0.140) | 0.19 (0.108)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.974417, ANCOVA; LS Mean Difference (Final Values) = -0.00, 95% CI 2-sided [-0.27 to 0.26]

40. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 16
Description: The CDLQI questionnaire is designed for use in children (4 to 16 years of age). It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses, and has a range of 0 to 30 (higher scores are indicative of greater impairment).
  LS Mean was calculated using MMRM model which includes treatment, baseline value, visit, the interaction of the baseline value-by-visit as covariates, the interaction of treatment by-visit, geographic region, age group, and baseline IGA (3 versus 4) score as fixed factors.
Time Frame: Baseline, Week 16
Population: All randomized, adolescent participants, with non-missing baseline CDLQI score, even if the participant does not take the assigned treatment, does not receive the correct treatment, or otherwise does not follow the protocol. One investigational site with eighteen participants was excluded from analysis due to GCP issues. MMRM was used to handle all missing data.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Lebrikizumab Q2W
Number analyzed (Participants) | 5 | 17
score on a scale | -3.4 (2.10) | -7.6 (1.13)
Statistical Analysis 1: Comparison: Placebo vs Lebrikizumab Q2W; Test type: Superiority; p = 0.084769, Mixed Models Analysis; LS Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-9.1 to 0.6]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: All randomized participants who received at least one dose of study drug. Gender specific events only occurring in male or female participants have had the number of participants at risk adjusted accordingly.
Groups:
- Induction - Lebrikizumab 250mg Q2W: Induction Period (Baseline-Week 16):
  500 milligram (mg) Lebrikizumab (2 x 250 mg) SC injections as a loading dose at Baseline and Week 2 visits followed by a single 250 mg Lebrikizumab injection Q2W from Week 4 until Week 14.
- Maintenance Blinded - Lebrikizumab Responder/ Placebo: Maintenance Period (Week 16 to Week 52): One 250 mg SC injection of Placebo Q2W.
- Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W: Maintenance Period (Week 16-Week 52):
  One 250 mg Lebrikizumab SC injection and one placebo SC injection as maintenance loading dose on Week 16 and two placebo SC injections on Week 18.
  One 250 mg Lebrikizumab SC injection Every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
- Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W: Maintenance Period (Week 16 to Week 52): One 250 mg Lebrikizumab SC injection Q2W.
- Maintenance Blinded - Placebo Responder/ Placebo: Maintenance Blinded - Placebo Responder/ Placebo
- Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W: Maintenance Period (Week 16 to Week 52):
  One 250 mg Lebrikizumab SC injection and one placebo SC injection as maintenance loading dose on Week 16 and two placebo SC injections on Week 18.
  One 250 mg Lebrikizumab SC injection Every 4 weeks (Q4W) on Weeks 20, 24, 28, 32, 36, 40, 44, and 48.
  One placebo SC injection Q4W on Weeks 22, 26, 30, 34, 38, 42, 46, and 50.
- Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W: Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W
- Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W: Maintenance Escape Period (Week 16 to Week 52): One 250 mg Lebrikizumab SC injection Q2W.
- Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W: Maintenance Escape Period (Week 16to Week 52): One 250 mg Lebrikizumab SC injection Q2W.
- Escape Arm Week 24 to 48 - Maintenance Lebrikizumab: Maintenance Escape Period (Week 24 to Week 48): One 250 mg Lebrikizumab SC injection Q2W.
Arm/Group | Induction - Placebo | Induction - Lebrikizumab 250mg Q2W | Maintenance Blinded - Lebrikizumab Responder/ Placebo | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W | Maintenance Blinded - Placebo Responder/ Placebo | Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W | Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W | Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W | Escape Arm Week 24 to 48 - Maintenance Lebrikizumab
All-Cause Mortality (participants affected / at risk) | 1/149 | 0/295 | 0/30 | 0/59 | 0/59 | 0/5 | 0/9 | 0/11 | 0/108 | 1/125 | 0/11
Serious Adverse Events (participants affected / at risk) | 4/149 | 2/295 | 1/30 | 0/59 | 2/59 | 0/5 | 2/9 | 0/11 | 1/108 | 5/125 | 0/11
Other Adverse Events (participants affected / at risk) | 97/149 | 157/295 | 15/30 | 32/59 | 36/59 | 3/5 | 4/9 | 8/11 | 68/108 | 77/125 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo (N=149) | Induction - Lebrikizumab 250mg Q2W (N=295) | Maintenance Blinded - Lebrikizumab Responder/ Placebo (N=30) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W (N=59) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W (N=59) | Maintenance Blinded - Placebo Responder/ Placebo (N=5) | Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W (N=9) | Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W (N=11) | Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W (N=108) | Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W (N=125) | Escape Arm Week 24 to 48 - Maintenance Lebrikizumab (N=11)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhegmatogenous retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paternal exposure during pregnancy (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/78 (1) | 0/147 (0) | 0/15 (0) | 0/34 (0) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Induction - Placebo (N=149) | Induction - Lebrikizumab 250mg Q2W (N=295) | Maintenance Blinded - Lebrikizumab Responder/ Placebo (N=30) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q4W (N=59) | Maintenance Blinded - Lebrikizumab Responder/Lebrikizumab Q2W (N=59) | Maintenance Blinded - Placebo Responder/ Placebo (N=5) | Maintenance Blinded - Placebo Responder/Lebrikizumab Q4W (N=9) | Maintenance Blinded - Placebo Responder/ Lebrikizumab Q2W (N=11) | Escape Arm Week 16 - Maintenance Open Label (OL) -Placebo Non-Responder/Lebrikizumab Q2W (N=108) | Escape Arm Week 16 - Maintenance OL- Lebrikizumab Non-Responder/Lebrikizumab Q2W (N=125) | Escape Arm Week 24 to 48 - Maintenance Lebrikizumab (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Auricular pseudocyst (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Paraesthesia ear (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atopic keratoconjunctivitis (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 2 (2) | 7 (7) | 1 (1) | 4 (6) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 12 (14) | 1 (1) | 0 (0)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Epiretinal membrane (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid erosion (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Keratoconus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst rupture (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vaccination site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to animal (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 21 (22) | 2 (3) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 3 (3) | 0 (0)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 6 (7) | 2 (2) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Demodicidosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis infected (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema herpeticum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema impetiginous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema infected (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes dermatitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Impetigo (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 15 (17) | 1 (2) | 3 (3) | 3 (5) | 0 (0) | 1 (1) | 2 (2) | 6 (10) | 10 (14) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 3 (3) | 4 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 3 (4) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Perineal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Superinfection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea barbae (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea capitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 5 (5) | 0 (0) | 3 (4) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (5) | 3 (3) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 1/78 (1) | 0/147 (0) | 0/15 (0) | 0/34 (0) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Accident at work (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injury corneal (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 4 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 2 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood alkaline phosphatase abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood testosterone decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte percentage decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mean cell haemoglobin concentration decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mean cell volume increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0/71 (0) | 0/148 (0) | 0/15 (0) | 0/25 (0) | 0/26 (0) | 0/2 (0) | 0/2 (0) | 0/5 (0) | 1/54 (1) | 0/70 (0) | 0/8 (0)
Urine ketone body present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/78 (0) | 0/147 (0) | 0/15 (0) | 0/34 (0) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 1/54 (1) | 0/55 (0) | 0/3 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 15 (17) | 1 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Narcolepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder due to general medical condition, insomnia type (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bladder disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0/78 (0) | 0/147 (0) | 0/15 (0) | 1/34 (3) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Bartholin's cyst (Reproductive system and breast disorders) | 0/78 (0) | 0/147 (0) | 0/15 (0) | 0/34 (0) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 1/54 (1) | 0/55 (0) | 0/3 (0)
Breast hyperplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast ulceration (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1/78 (1) | 0/147 (0) | 0/15 (0) | 0/34 (0) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0/78 (0) | 0/147 (0) | 0/15 (0) | 1/34 (1) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Penis disorder (Reproductive system and breast disorders) | 0/71 (0) | 0/148 (0) | 0/15 (0) | 0/25 (0) | 0/26 (0) | 0/2 (0) | 0/2 (0) | 0/5 (0) | 0/54 (0) | 1/70 (1) | 0/8 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0/78 (0) | 0/147 (0) | 0/15 (0) | 0/34 (0) | 1/33 (1) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0/78 (0) | 1/147 (1) | 0/15 (0) | 0/34 (0) | 0/33 (0) | 0/3 (0) | 0/7 (0) | 0/6 (0) | 0/54 (0) | 0/55 (0) | 0/3 (0)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Alopecia areata (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 38 (41) | 27 (31) | 3 (3) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 6 (8) | 2 (2)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diffuse alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hair disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin lesion inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
One investigational site with eighteen participants was excluded from analysis due to GCP issues.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/67/NCT04178967/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04178967/SAP_001.pdf